CLINICAL TRIAL: NCT07076914
Title: Prophylactic Proton Pump Inhibition for Esophageal Protection in Lung Radiation Therapy: A Randomized Clinical Trial
Brief Title: Prophylactic Proton Pump Inhibition for Esophageal Protection in Lung Radiation Therapy
Acronym: PPI-PROTECT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPI-PROTECT
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Primary Lung Cancer; Non Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: proton pump inhibitor; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Proton Pump Inhibitors; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Radiation delivered as per standard institutional approaches
- Prophylactic Proton Pump Inhibitor (Experimental): Daily use of pantoprazole magnesium, rabeprazole or lansoprazole
  Interventions: Drug: Experimental (Health Canada Approved Proton Pump Inhibitors)

INTERVENTIONS:
Drug: Experimental (Health Canada Approved Proton Pump Inhibitors) — The intervention uses a proton pump inhibitor as a preventative measure
  Other Names: Proton Pump Inhibitor; Pantoprazole magnesium; rabeprazole
  Arms: Prophylactic Proton Pump Inhibitor

SUMMARY:
A randomized controlled trial to assess the impact of prophylactic proton pump inhibitor use to improve esophagitis in lung cancer patients undergoing radiation. Patients will be randomized into a standard of care arm or the prophylactic proton pump (daily) arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

  * Willing to provide informed consent
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-3
  * Life expectancy of at least 3 months
  * Primary lung malignancy of any stage (including NSCLC and small cell lung cancer). Histologic/pathologic diagnosis is preferred, but not required.
  * Receiving a prescribed dose of at least 40 Gy in 15 fractions (or equivalent). Eligible fractionations include, but are not limited to, 60 Gy in 30 fractions, 55 Gy in 20 fractions, and 40-45 Gy in 15 fractions.
  * On radiation planning, at least 5 cc of esophagus is receiving at least 95% of prescription dose

Exclusion Criteria:

* • Serious medical comorbidities precluding radiotherapy

  * Use of PPI within 3 months prior to enrollment
  * Allergy to PPI
  * Odynophagia (painful swallowing) prior to enrollment
  * Pregnant or lactating women

Note: previous radiation to the thorax is allowed, as long as the composite plan of current and prior radiation doses meet standard institutional dose constraints, in the opinion of the treating radiation oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2032-10-02 (Estimated)

PRIMARY OUTCOMES:
Worst patient-reported esophageal pain score during radiation | baseline last week of radiation post-treatment
  Assessed with the 11-Numeric Rating Scale using weekly questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No